CLINICAL TRIAL: NCT05502406
Title: Effectiveness of Manual Myofascial Release Versus Instrument Assisted Soft Tissue Mobilization (IASTM) in Patients With Chronic Neck Pain"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2022/9
Record Dates: First submitted 2022-08-10; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Chronic Neck Pain

STUDY DESIGN:
Intervention Model Description: compare two treatment techniques the study type will be parallel experimental study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IASTM (Experimental): The participants of the respective group will receive myofascial release using a C shaped glider, by the help of gentle horizontal strokes the targeted soft tissue restrictions will be relieved over the cervicodorsal fascia
  Interventions: Procedure: Instrument Assisted Soft tissue Mobilization
- MMFR (Experimental): The participants of the respective group will recieve manual soft tissue release over the cervicodorsal fascia using velvet glove technique for a period of 5 to 7 mins inorder to set free any adhesion in the underlying myofascia
  Interventions: Procedure: Manual Myofascial Release

INTERVENTIONS:
Procedure: Instrument Assisted Soft tissue Mobilization — Using a C shaped IASTM tool gentle horizontal stroking at an angle of 45 degree will be given over the cervicodorsal fascia
  Arms: IASTM
Procedure: Manual Myofascial Release — Participants will receive myofascial release through velvet glove technique on upper trapezius and sternocleidomastoid muscle using four strokes in the following fashion:
  * Begin superior to the clavicle with a loose fist and move the back of the hand over the upper trapezius, fastening the tissue and bringing it over the table.
  * The next stroke addresses the curve of the neck, again hooking the tissue while moving the bak of your fist towards the table.
  The last stroke goes over the entire cervical spine hooking over the sternocleidomastoid muscle bringing it into myofascial release. Stay away from the carotid pulse, and incase a pulse is felt, do not apply pressure and reposition your hand
  Arms: MMFR

SUMMARY:
Neck pain has a global prevalence of 30%, being the fourth leading cause of disability among general population and is more prevalent among females than males, as per concluded by evidence. It is undoubtedly the need of time, to address its proper treatment and to hinder its recurrence amongst the general population. The current physical therapy management of neck pain is more focused towards achieving the short term goals for the patient rather than addressing and amending the actual cause of its relapse. Manual Myofascial Release is one of the very effective treatment used to release soft tissue and fascial adhesions over the myofascia inorder to relieve chronic neck pain. The study aims to compare this manual treatment against Instrument Assisted soft tissue mobilization in order to determine which of the two provides improved outcome in terms of pain, neck disability and cervical Range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female participants belonging to the age group of 18 to 40 years
* Participants suffering from neck pain for more than 3months.

Exclusion Criteria:

* Recent history of Whiplash Injury.
* Recent traumatic history of head, cervical spine, shoulder girdle or fractures of the cervical spine or shoulder complex.
* History of Cervical Radiculopathy, spondylosis, spondylolisthesis, disc prolapse, any other systemic disease or vascular syndrome such as vertebro-basilar Insufficiency.
* Diagnosed Fibromyalgia, myopathy or myelopathy
* Sensory/Motor dysfunction owing to any neurological pathology in the mid or upper back.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 2 weeks
  Pain will be measured using numeric pain rating scale which is a 10 point scale characterising 0 as no pain and 10 as worst possible pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Punjab Province, Pakistan